CLINICAL TRIAL: NCT02043444
Title: Comparison of FDG PET-CT Estimated Testis Functional Value Between Patients Having Positive Testicular Sperm Cells Extraction and Patients With a Negative Extraction, in Men With Azoospermia
Brief Title: Secretory Azoospermia and FDG (Fluoro Deoxyglucose) PET-CT
Acronym: AzoPredHisto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12 555 01; PHRC 2012 (Other Grant/Funding Number: PHRC)
Record Dates: First submitted 2013-12-13; First posted 2014-01-23 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2020-11

CONDITIONS: Fertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- secretory azoospermia (Experimental): 110 men with secretory azoospermia will have FDG PET-CT
  Interventions: Radiation: FDG PET-CT
- excretory azoospermia (Active Comparator): 30 men with secretory azoospermia will have FDG PET-CT
  Interventions: Radiation: FDG PET-CT
- normospermia (Placebo Comparator): 20 men with secretory azoospermia will have FDG PET-CT
  Interventions: Radiation: FDG PET-CT

INTERVENTIONS:
Radiation: FDG PET-CT

SUMMARY:
Compare FDG PET-CT parameters between azoospermia patients having an extraction of sperm cells by positive testicular extraction and those with a negative extraction.

DETAILED DESCRIPTION:
One third of infertilities is of exclusive male origin and one third of mixed origin (presence of a male factor). Ten percent of infertile male have azoospermia with a secretory origin in most of cases. Surgical extraction of spermatozoa from testicle is the unique possibility to increase the chance for these men to have children using in vitro fecundation. However, surgical extraction of spermatozoa is successful in 50% of these patients. To date, none of the methods for exploration of male fertility (spermogram, hormonal investigation - with dosage of FSH (follicle stimulating hormone) and inhibin B - and scrotal ultrasound) can predict the success of surgical sperm cells extraction. We also miss the prognostic markers of the testicular function recovery after sterilizing treatments (chemotherapy, radiotherapy). The presence of GLUT3 (glucose) transporters, which are responsible for the fluoro deoxyglucose uptake, has been reported in seminiferous tubules. We have previously shown in a pilot study on a population of men without testis cancer that FDG PET-CT parameters - including the standardized uptake value mean, the standardized uptake value max, and the functional testicular volume - were correlated with the parameters of spermogram (sperm count, motility, vitality). These findings open the way to investigations on the role of the FDG PET-CT in evaluation of secretory azoospermia.

ELIGIBILITY:
Inclusion Criteria:

absence of sperm cells on 2 spermograms in 3 months interval testicular size has to be determined in order to categorized in a group to accept surgery-

Exclusion Criteria:

allergy to fluoro deoxyglucose clinical varicocele

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
measure of standardized uptake value (SUV) | 1 month

SECONDARY OUTCOMES:
comparison between functional volume with PET exam and volume obtained by scrotal echography | 1 month

OTHER OUTCOMES:
comparison functional volume with FSH and inhibin | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Eric HUYGHE, MD, Principal Investigator — University Hospital, Toulouse
Locations (5):
- France (5):
  - UHBordeaux, Bordeaux
  - University Hospital, Lille
  - Centre européen Georges Pompidou, Paris
  - University Hospital, Rouen
  - UHToulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferretti L, Sargos P, Gross-Goupil M, Izard V, Wallerand H, Huyghe E, Rigot JM, Durand X, Benoit G, Ferriere JM, Droupy S. Testicular-sparing surgery for bilateral or monorchide testicular tumours: a multicenter study of long-term oncological and functional results. BJU Int. 2014 Dec;114(6):860-4. doi: 10.1111/bju.12549. Epub 2014 Aug 16. PMID 24180380
- [Result] Dierickx LO, Bettiol C, Huglo D, Marcelli F, Sibert L, Gouel P, Ferretti L, Orlhac F, Huyghe E. Is 18F-fluorodexyglucose testicular uptake using positron emission tomography/computed tomography correlated with the results of a testicular sperm extraction procedure in the case of azoospermia (French prospective multicenter AZOPREDHISTOTEP study)? Eur J Nucl Med Mol Imaging. 2025 Nov 21. doi: 10.1007/s00259-025-07583-7. Online ahead of print. PMID 41269291